CLINICAL TRIAL: NCT03123549
Title: Clinical Study Protocol for the Investigation Of The Two Level Simplify® Cervical Artificial Disc
Brief Title: Investigation of the Two Level Simplify® Cervical Artificial Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G150206
Record Dates: First submitted 2017-03-29; First posted 2017-04-21 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Degenerative Disc Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Simplify Disc (Experimental): Simplify Disc at two levels of the cervical spine
  Interventions: Device: Simplify Disc
- Historical Control (No Intervention): This study will utilize a non-concurrent historical control with subject-level data on a parallel group design. The historical control group will be formed from the randomized ACDF arm of a previously completed two level cervical disc trial.

INTERVENTIONS:
Device: Simplify Disc — Simplify Disc at two levels of the cervical spine
  Arms: Simplify Disc

SUMMARY:
This study is intended to demonstrate that the Simplify® Cervical Artificial Disc (Simplify® Disc) is at least as safe and effective as conventional anterior cervical discectomy and fusion (ACDF) when used to treat two contiguous discs from C3 to C7 following discectomy at two contiguous levels for intractable radiculopathy (arm pain and/or a neurological deficit) with neck pain or myelopathy due to abnormalities localized to the levels of the two contiguous disc spaces in subjects who are unresponsive to conservative management.

DETAILED DESCRIPTION:
The objective of this clinical study is to evaluate the safety and effectiveness of the two-level Simplify® Disc compared to conventional two-level ACDF in skeletally mature patients for reconstruction of two contiguous discs from C3 to C7 following discectomy at two contiguous levels for intractable radiculopathy (arm pain and/or a neurological deficit) with neck pain or myelopathy due to abnormalities localized to the levels of the two contiguous disc spaces that are unresponsive to conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Has cervical degenerative disc disease at two (2) adjacent cervical levels (from C3 C7) requiring surgical treatment and involving intractable radiculopathy, myelopathy, or both;
* Has a herniated disc and/or osteophyte formation at each level to be treated that is producing symptomatic nerve root and/or spinal cord compression. The condition is documented by patient history (e.g., neck pain with arm pain, functional deficit and/or neurological deficit), and the requirement for surgical treatment is evidenced by radiographic studies (e.g., CT, MRI, x-rays, etc.);
* Has been unresponsive to non-operative treatment for at least six weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management;
* Has no previous surgical intervention at the involved levels or any subsequent planned/staged surgical procedure at the involved or adjacent level(s);
* Must be at least 18 years of age and be skeletally mature at the time of surgery;
* Has a preoperative Neck Disability Index (NDI) ≥ 30;
* Has a preoperative neck pain score > 8 based on the preoperative Neck and Arm Pain Questionnaire;
* If a female of childbearing potential, patient is non-pregnant, non-nursing, and agrees not to become pregnant during the study period;
* Is willing to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

* Has a cervical spinal condition other than symptomatic cervical DDD requiring surgical treatment at the involved levels;
* Has documented or diagnosed cervical instability relative to adjacent segments at either level, defined by dynamic (flexion/extension) radiographs showing:

  * Sagittal plane translation > 3.5 mm, or
  * Sagittal plane angulation > 20°;
* Has more than two cervical levels requiring surgical treatment;
* Has a fused level (or artificial disc replacement) adjacent to the levels to be treated;
* Has severe pathology of the facet joints of the involved vertebral bodies;
* Has had previous surgical intervention at either one or both of the involved levels or at adjacent levels;
* Axial neck pain only (no radicular or myelopathy symptoms);
* Has been previously diagnosed with osteopenia or osteomalacia;
* Has any of the following that may be associated with a diagnosis of osteoporosis (if "Yes" to any of the below risk factors, a DEXA Scan will be required to determine eligibility):

  * Postmenopausal non-black female over 60 years of age who weighs less than 140 pounds;
  * Postmenopausal female who has sustained a non-traumatic hip, spine, or wrist fracture;
  * Male over the age of 70;
  * Male over the age of 60 who has sustained a non-traumatic hip or spine fracture.
  * If the level of bone mineral density is a T score of -1.5 or lower (i.e., -1.6, 1.7, etc.), then the patient is excluded from the study
* Has presence of spinal metastases;
* Has overt or active bacterial infection, either local or systemic;
* Has insulin-dependent diabetes;
* Has chronic or acute renal failure or prior history of renal disease;
* Known PEEK, ceramic, titanium allergy;
* Is mentally incompetent (if questionable, obtain psychiatric consult);
* Is a prisoner;
* Is pregnant;
* Is currently an alcohol and/or drug abuser or currently undergoing treatment for alcohol and/or drug abuse;
* Is involved with current or pending litigation regarding a spinal condition;
* Has received drugs that may interfere with bone metabolism within two weeks prior to the planned date of spinal surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs;
* Has a history of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers-Danlos Syndrome, or osteogenesis imperfecta);
* Has a condition that requires postoperative medications that interfere with the stability of the implant, such as steroids. (This does not include low-dose aspirin for prophylactic anticoagulation and routine perioperative anti-inflammatory drugs);
* Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, Study Director — NuVasive
Locations (18):
- United States (18):
  - Orthopaedic Education and Research Institute of Southern California, Orange, California
  - The Spine Institute for Spine Restoration, Santa Monica, California
  - Spine Education and Research Foundation, Thornton, Colorado
  - Connecticut Orthopaedic Specialists, Hamden, Connecticut
  - Kennedy-White orthopedic Center, Sarasota, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine institute of Louisiana, Shreveport, Louisiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - Buffalo Spine Surgery, Lockport, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Oregon Neurosurgery, Springfield, Oregon
  - Texas Spine Consultants, Addison, Texas
  - Texas Back Institute, Plano, Texas
  - The Disc Replacement Center, West Jordan, Utah
  - Virginia Spine Institute, Reston, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Simplify Medical Website for the Simplify Disc Trial — http://www.simplifymedical.com/simplify-disc/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical control was used for control arm. The only subjects enrolled under this study were investigational subjects (Simplify Disc).
Groups:
- Historical Control - Anterior Cervical Discectomy and Fusion (ACDF): This study will utilize a non-concurrent historical control with subject-level data on a parallel group design. The historical control group will be formed from the randomized ACDF arm of a previously completed two level cervical disc trial.
Period: Overall Study
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Started | 182 | 170
Completed | 168 (For subject accounting purposes, "completed" is defined as having either a 24-month change in NDI score or an available motor neurological assessment at 24-months.) | 127 (For subject accounting purposes, "completed" is defined as having either a 24-month change in NDI score or an available motor neurological assessment at 24-months.)
Not Completed | 14 | 43

BASELINE CHARACTERISTICS:
Population: One hundred eighty-two (182) subjects were enrolled in the Simplify® Cervical Artificial Disc analysis population. An additional 18 Simplify® Cervical Artificial Disc subjects were training subjects and were not included in the analysis. The historical ACDF control analysis population included 170 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simplify Disc | Historical Control | Total
Number analyzed (Participants) | 182 | 170 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.25 (9.39) | 47.45 (7.89) | 48.38 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 184
  Male | 87 | 81 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data not captured for historical control group.
  Participants
    number analyzed (Participants) | 182 | 0 | 182
    Hispanic or Latino | 5 |  | 5
    Not Hispanic or Latino | 177 |  | 177
    Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 170 | 157 | 327
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 182 | 170 | 352

OUTCOME MEASURES:

1. Primary Outcome: Composite Clinical Success (CCS) Rate of the Simplify® Disc
Description: Individual success is defined as at least a 15 point improvement in Neck Disability Index (NDI) Score at 24 months compared with baseline, maintenance or improvement in neurologic status at 24 months compared with baseline, no additional surgical procedure at the index level within 24 months, and the absence of a serious adverse event classified as implant-associated or implant/surgical procedure-associated within 24 months.
  NDI scale is reported in a range from 0 - 100, with 0 consistent with best ability to function and 100 with worst ability to function.
Time Frame: 24 Months
Population: While 168 Simplify Disc subjects and 127 historical control subjects were considered completers for subject accounting purposes, 173 (Simplify Disc) and 145 (ACDF) subjects were evaluable for composite clinical success. This is due to the fact that some subjects were known failures prior to the 24-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control
Number analyzed (Participants) | 173 | 145
Participants | 153 | 105
Statistical Analysis 1: Comparison: Simplify Disc vs Historical Control; Test type: Superiority; p = 0.017, t-test, 1 sided

2. Secondary Outcome: Neurological Status
Description: Neurological success was defined as maintenance or improvement in neurologic status at Month 24 as compared to baseline, as determined by the independent Clinical Events Committee (CEC). The CEC reviews neurological exams of motor, sensory, reflex, and myelopathic gait to make an adjudication determination.
Time Frame: Baseline, 24mos
Population: While 127 historical control subjects were considered completers for subject accounting purposes, 128 historical subjects had sufficient neurological data available for CEC determination of maintenance or improvement of neurological status.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 168 | 128
Participants
  Improved | 140 | 106
  Maintained | 28 | 19
  Deteriorated | 0 | 3

3. Secondary Outcome: Number of Subjects With 15-point Improvement in NDI at 3 Months (Time to Recovery)
Description: Time to recovery is defined as time to first 15-point improvement in NDI NDI scale is reported in a range from 0 - 100, with 0 consistent with best ability to function and 100 with worst ability to function.
Time Frame: Baseline, 3mos
Population: While 168 Simplify Disc subjects and 127 historical control subjects were considered completers for subject accounting purposes at 24 months, 177 (Simplify Disc) and 154 (ACDF) subjects had evaluable change in NDI scores at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 177 | 154
Participants
  15-Point Improvement (Yes) | 160 | 123
  15-Point Improvement (No) | 17 | 31

4. Secondary Outcome: Neck Pain Intensity Questionnaire
Description: Changes of at least 2 points on a 10-point scale will be regarded as clinically significant (0=no pain; 10=worst pain)
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 158 Simplify Disc subjects had change in Neck Pain Intensity data at 24 months due to missed questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 158 | 127
Participants
  Success | 147 | 110
  Fail | 11 | 17

5. Secondary Outcome: Arm Pain Intensity Questionnaire
Description: Changes of at least 2 points on a 10-point scale will be regarded as clinically significant (0=no pain; 10=worst pain)
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 158 Simplify Disc subjects had change in Arm Pain Intensity data at 24 months due to missed questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 158 | 127
Participants
  Success | 142 | 108
  Failure | 16 | 19

6. Secondary Outcome: Patient Questionnaires- Treatment Satisfaction Survey
Description: Question 1 - "I am satisfied with the results of my surgery" was compared between groups at Month 24. Answer options ranged from definitely true to definitely false.
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects and 127 historical control subjects were considered completers for subject accounting purposes, 172 (Simplify Disc) and 145 (ACDF) subjects had evaluable treatment satisfaction data at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 172 | 145
Participants
  Definitely true | 131 | 99
  Mostly true | 26 | 30
  Don't know | 8 | 7
  Mostly false | 5 | 4
  Definitely false | 2 | 5

7. Secondary Outcome: SF-36v2 Health Survey Physical Component Score (PCS) Maintenance or Improvement
Description: The PCS is a sub-score of the SF-36. The SF-36 is a multipurpose survey with 36 questions. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related quality-of-life. Higher scores indicate better outcomes. Scores range from 0-50. Maintenance or improvement was defined as PCS(Postop) - PCS(Preop) ≥0.
Time Frame: Baseline, 24mos
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 158 Simplify Disc subjects had SF-36 data available at 24 months due to missed questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 158 | 127
Participants
  Maintenance or improvement | 146 | 114
  Absence of maintenance or improvement | 12 | 13

8. Secondary Outcome: SF-36 Mental Component Score (MCS) Maintenance or Improvement
Description: The MCS is a sub-score of the SF-36. The SF-36 is a multipurpose survey with 36 questions. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related quality-of-life. Higher scores indicate better outcomes. Scores range from 0-50. Maintenance or improvement was defined as MCS(Postop) - MCS(Preop) ≥0.
Time Frame: Baseline, 24mos.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 158 | 127
Participants
  Maintenance or improvement | 125 | 94
  Absence of maintenance or improvement | 33 | 33

9. Secondary Outcome: Dysphagia Handicap Index (DHI)
Description: Dysphagia Handicap Index (DHI scale) for the investigational Simplify® Disc at 24 months compared to baseline. A higher score is indicative of a less desirable outcome. It is scored 0-100.
  Data was not collected on DHI in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24mos.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simplify Disc
Number analyzed (Participants) | 167
score on a scale | 6.9 (10.7)

10. Secondary Outcome: Physician's Perception of Results
Description: Results at 24 months for the investigational Simplify® Disc and at 24 months for the control ACDF will also be categorized by the physician according to their perception of the results. Available responses include excellent, good, fair, and poor. Maintenance or improvement was defined as either maintenance of the assigned preoperative grade or any shift to a more favorable grade postoperatively (e.g. poor to fair, fair to good).
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects and 127 historical control subjects were considered completers for subject accounting purposes, 170 (Simplify Disc) and 145 (ACDF) subjects had evaluable Physician's Perception of Results data at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
Number analyzed (Participants) | 170 | 145
Participants
  Excellent | 139 | 85
  Good | 26 | 42
  Fair | 3 | 15
  Poor | 2 | 3

11. Secondary Outcome: Change in Average Disc Height (Superior Index Level)
Description: Average disc height (superior index level) at 24 months was compared to the baseline measurement and the change was calculated. Measurements were scored by an independent core lab. Average disc height is calculated as the simple average of the anterior and posterior disc heights.
  Data was not collected on disc height in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 164 Simplify Disc subjects had evaluable radiographs for this assessment at 24 months due to missed x-rays or poor image quality which limited analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Simplify Disc
Number analyzed (Participants) | 164
mm | 1.19 (0.81)

12. Secondary Outcome: Change in Average Disc Height (Inferior Index Level)
Description: Average disc height (inferior index level) at 24 months was compared to the baseline measurement and the change was calculated. Measurements were scored by an independent core lab. Average disc height is calculated as the simple average of the anterior and posterior disc heights.
  Data was not collected on disc height in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24M
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 157 Simplify Disc subjects had evaluable radiographs for this assessment at 24 months due to missed x-rays or poor image quality which limited analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Simplify Disc
Number analyzed (Participants) | 157
mm | 0.84 (0.96)

13. Secondary Outcome: Superior Adjacent Level Disc Degeneration (ALDD)
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) above the index level based on X-ray images. Degeneration was graded as none (no degenerative changes), doubtful (Minimal osteophytosis only), minimal (Definite osteophytosis with some sclerosis of anterior part of vertebral plates), moderate (Marked osteophytosis and sclerosis of vertebral plates with slight narrowing of disk space), severe (Large osteophytes, marked sclerosis of vertebral plates, and marked narrowing of disk space), indeterminate, or unable to assess.
  Data was not collected on ALDD in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 166 Simplify Disc subjects had evaluable radiographs for this assessment at 24 months due to missed x-rays or poor image quality which limited analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 166
Participants
  None | 100
  Doubtful | 45
  Minimal | 16
  Moderate | 2
  Severe | 1
  Indeterminate | 0
  Unable to assess | 2

14. Secondary Outcome: Inferior Adjacent Level Disc Degeneration (ALDD)
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) below the index level based on X-ray images. Degeneration was graded as none (no degenerative changes), doubtful (Minimal osteophytosis only), minimal (Definite osteophytosis with some sclerosis of anterior part of vertebral plates), moderate (Marked osteophytosis and sclerosis of vertebral plates with slight narrowing of disk space), severe (Large osteophytes, marked sclerosis of vertebral plates, and marked narrowing of disk space), indeterminate, or unable to assess.
  Data was not collected on ALDD in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24mos.
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 166
Participants
  None | 110
  Doubtful | 20
  Minimal | 9
  Moderate | 2
  Severe | 1
  Indeterminate | 21
  Unable to assess | 3

15. Secondary Outcome: Facet Degeneration (Superior Index Level)
Description: Facet degeneration was assessed using MRI for the investigational Simplify Disc at 24 months compared to baseline. Degeneration was graded as none (normal facet joint space), mild (narrowing of the facet joint space and / or small osteophytes and / or mild hypertrophy of the articular process), moderate (narrowing of the facet joint space and/or moderate osteophytes and/or moderate hypertrophy of the articular process and / or mild subarticular bone erosions), severe (Narrowing of the facet joint space and/or large osteophytes and/or severe hypertrophy of the articular process and/or severe subarticular bone erosions and/or subchondral cysts), indeterminate, or unable to assess.
  Facet degeneration was not assessed in the ACDF historical control group, as there is no 24 month MRI. This was pre-specified in the study design.
Time Frame: Baseline, 24mos.
Population: While 168 Simplify Disc subjects were considered completers for subject accounting purposes, 166 Simplify Disc subjects had an evaluable MRI for this assessment at 24 months due to missed MRIs.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 166
Participants
  None | 87
  Mild | 64
  Moderate | 13
  Severe | 0
  Indeterminate | 0
  Unable to assess | 2

16. Secondary Outcome: Facet Degeneration (Inferior Index Level)
Description: as for outcome 15
Time Frame: Baseline, 24mos.
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 166
Participants
  None | 96
  Mild | 60
  Moderate | 8
  Severe | 0
  Indeterminate | 0
  Unable to assess | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected continuously throughout study follow-up period. Results are reported through study day 790.
Groups:
- Historical Control - Anterior Cervical Discectomy and Fusion (ACDF): This study will utilize a non-concurrent historical control with subject-level data on a parallel group design. The historical control group will be formed from the randomized ACDF arm (N=188) of a previously completed two level cervical disc trial.
Arm/Group | Simplify Disc | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF)
All-Cause Mortality (participants affected / at risk) | 2/182 | 1/170
Serious Adverse Events (participants affected / at risk) | 32/182 | 62/170
Other Adverse Events (participants affected / at risk) | 96/182 | 145/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=182) | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF) (N=170)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Infection (all other infections-NOT at cervical surgical site) (Infections and infestations) | 6 (7) | 2 (2)
Hematoma or seroma (Vascular disorders) | 2 (2) | 0 (0)
Accidental trauma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Low back pain (no narcotic given) (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Appendicular arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
Cervical Radiculopathy (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Lumbar Radiculopathy (Musculoskeletal and connective tissue disorders) | 8 (8) | 13 (14)
Pain (no narcotic given) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal complications including ileus, nausea and vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Blood loss (greater than 500ml) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Difficulty with urination (Renal and urinary disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Development of DDD at adjacent levels (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dural injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychological Illness (Psychiatric disorders) | 0 (0) | 2 (2)
Soft tissue damage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis/Skin allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Low back pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Nonunion/pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
Inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Implant collapse or subsidence (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spondylosis acquista (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Other (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac Event (Cardiac disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=182) | Historical Control - Anterior Cervical Discectomy and Fusion (ACDF) (N=170)
Infection (all other infections-NOT at cervical surgical site) (Infections and infestations) | 10 (12) | 18 (20)
Accidental trauma (Injury, poisoning and procedural complications) | 18 (20) | 37 (42)
Dermatitis/Skin allergy (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (9)
Low back pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (11)
Appendicular arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 25 (30)
Cervical Radiculopathy (Musculoskeletal and connective tissue disorders) | 22 (26) | 31 (34)
Inflammation (Musculoskeletal and connective tissue disorders) | 21 (23) | 30 (34)
Lumbar Radiculopathy (Musculoskeletal and connective tissue disorders) | 18 (18) | 16 (16)
Numbness - increased from pre-op or prior visit (Nervous system disorders) | 4 (4) | 14 (14)
Pain (no narcotic given) (Musculoskeletal and connective tissue disorders) | 22 (24) | 34 (38)
Compressive Neuropathy (Nervous system disorders) | 12 (12) | 18 (18)
Gastrointestinal complications including ileus, nausea and vomiting (Gastrointestinal disorders) | 5 (5) | 12 (17)
Development of DDD at adjacent levels (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 14 (14)
Headache (Nervous system disorders) | 9 (9) | 23 (24)
Pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 5 (5) | 12 (12)
Spasm (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (13)
Neck Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9)

LIMITATIONS AND CAVEATS:
ACDF data is presented as a historical control fusion group from a previously completed IDE trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03123549/Prot_SAP_000.pdf